CLINICAL TRIAL: NCT01666821
Title: A Population-based Study of Macular Choroidal Neovascularization Using Optical Coherence Tomography in a Chinese Population
Brief Title: A Population-based Study of Macular Choroidal Neovascularization in a Chinese Population
Status: Completed | Type: Observational
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jun Hu, Department of ophthalmology, Shuguang hospital(Baoshan branch),Shanghai University of TCM, Shanghai University of Traditional Chinese Medicine
Other Study IDs: 04-E-1
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Geographic Atrophy; Wet Macular Degeneration; Retinal Drusen
Keywords: macular degeneration; choroidal neovascularization
MeSH Terms: conditions — Geographic Atrophy; Wet Macular Degeneration; Retinal Drusen; Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- early and intermediate-stage AMD: Follow-up observation was implemented in whose fundus examination show lesions in the early and intermediate-stage AMD
  Interventions: Other: Follow-up observation

INTERVENTIONS:
Other: Follow-up observation — a epidemiologic survey of ocular diseases in an adult population (>45 years old) in Youyi Street, Baoshan District, Shanghai, China, conducted to determine the prevalence of AMD in the region. To this end, we utilized routine ocular examinations

SUMMARY:
To investigate pathomorphological and functional variations of choroidal neovascularization (CNV) in age-related macular degeneration (AMD) in a Chinese population using optical coherence tomography (OCT) to find which kinds of Fundus characteristics indicated exudative AMD.

DETAILED DESCRIPTION:
This population-based study enrolled 59 patients (>45 years old; 70 eyes) with early and intermediate-stage AMD from Youyi Street, Baoshan District, Shanghai, China. Comprehensive standardized ophthalmic examinations included visual acuity, anterior segment analysis by slit lamp, dilated fundus evaluation by direct ophthalmoscopy, 90D handheld lens, fundus photography, fluorescein angiography (FFA), and fast optic disk scans using OCT. The macular CNV characteristic profiles in early and intermediate-stage AMD were determined by OCT. Data were obtained at first visit and 6 to 24 months follow-up, and FFA and OCT outcomes of early and intermediate-stage AMD patients were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* adults citizens aged above 45 years

Exclusion Criteria:

* lost samples

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: recruited 1813 adults citizens aged above 45 years by probability sampling from the Youyi Street, Baoshan District, Shanghai, China for an epidemiologic survey. All participants gave written informed consent, and this study was approved by the local Ethics Committee in accordance with the Helsinki Declaration.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2004-05; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
change of the early and intermediate-stage AMD | May 2004-September 2008
  Drusen with unclear boundaries and obvious pigment proliferation, with hypofluorescence around drusens seen on FFA and a slight small arch field located in the retinal pigment epithelium (RPE)/choriocapillary layer (CCL) on OCT indicated exudative AMD.

CONTACTS AND LOCATIONS:
Overall Officials: zhao jie, master, Principal Investigator — Director of ophthalmology
Locations (1):
- Youyi Street, Shanghai, Baoshan District, China